CLINICAL TRIAL: NCT06027788
Title: Embolic Protection in Patients Undergoing High-Risk Valve Surgery
Brief Title: CTSN Embolic Protection Trial
Acronym: EMPRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Annetine Gelijns, Professor of Health Policy, Chair Department of Health Evidence & Policy, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY-23-00417; 5U01HL088942-16 (NIH)
Record Dates: First submitted 2023-08-21; First posted 2023-09-07 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Delirium; Ischemic Stroke; Acute Kidney Injury; Heart Valve Disease; Coronary Artery Disease
Keywords: Embolic Protection; Cardiac Surgery; CardioGard
MeSH Terms: conditions — Delirium; Ischemic Stroke; Acute Kidney Injury; Heart Valve Diseases; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to the embolic protection device or to a standard cannula in the OR immediately after sternotomy and confirmation by the surgical team of the patient's suitability for the proposed intervention (CardioGard embolic protection device).
Who Masked: Outcomes Assessor
Masking Description: The nature of the study precludes masking surgeons from treatment assignment. Investigators will, however, be blinded to all data from other clinical sites, except serious unexpected adverse events possibly or probably related to the intervention for Institutional Review Board (IRB)/Research Ethics Board (REB) reporting purposes. Patients will be blinded as to treatment assignment. All neurocognitive scoring and delirium assessments will be analyzed by neurocognitive core laboratory personnel who will be blinded to treatment assignment and clinical outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CardioGard Embolic Protection Cannula (Active Comparator): In patients assigned to the embolic protection device group, the CardioGard Embolic Protection Cannula is used instead, according to the manufacturer's instructions for use (IFU).
  Interventions: Device: CardioGard Embolic Protection Cannula
- Standard Aortic Cannula (Placebo Comparator): In patients assigned to the standard cannula group, standard cannulation techniques are performed using any standard aortic cannula of the surgeon's choice
  Interventions: Device: Standard Aortic Cannula

INTERVENTIONS:
Device: CardioGard Embolic Protection Cannula — The CardioGard embolic protection cannula is a device that combines the function of a standard aortic cannula with an added suction mechanism to capture debris that may result from cardiac surgery. The device is comprised of 2 hollow tubes. The first tube is the standard main forward-flow tube to return oxygenated blood to the patient's aorta. The second tube attached to an existing bypass vent port, is a novel element located posteriorly to the main tube; its function is to facilitate blood and particle suction by directing the blood back to the reservoir of the coronary bypass machine, while the retrieved embolic debris is eliminated through the filter of the venous reservoir.
  Arms: CardioGard Embolic Protection Cannula
Device: Standard Aortic Cannula — An aortic cannula is a device that is used routinely during cardiac surgery to return oxygenated blood from the cardiac bypass machine into the patient's aorta.
  Arms: Standard Aortic Cannula

SUMMARY:
This is a prospective, multi-center, randomized effectiveness trial of the CardioGard Embolic Protection Cannula in high-risk valve surgery patients.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled clinical trial that will evaluate the effectiveness and safety of the CardioGard embolic protection cannula compared to a standard cannula. The enrollment period is expected to last 30 months, and all patients will be followed for 12 months post procedure.

RANDOMIZATION Patients will be randomized 1:1 to the embolic protection device or to a standard cannula in the operating room (OR) immediately after sternotomy and confirmation by the surgical team of the patient's suitability for the proposed intervention (CardioGard embolic protection device). Randomization will be with equal allocation and stratified by site and by procedure (i.e., isolated valve surgery or combined procedures, such as double valve or valve plus coronary artery bypass grafting, CABG). The randomization assignment will be controlled centrally and performed through a web-based data collection system that automates the delivery of the randomization codes. From the point of treatment assignment, primary efficacy will be analyzed by intention-to-treat; that is, the patients will be grouped by their assignments at randomization regardless of whether or not they actually received the treatment to which they were assigned.

STUDY POPULATION The patient population for this trial consists of patients age ≥ 60 undergoing different types of valve surgery with or without CABG via full or minimal-access sternotomy using legally marketed valve(s). Specific inclusion and exclusion criteria are listed below. All patients who meet the eligibility criteria may be included in the study regardless of gender, race, or ethnicity.

SUBSTUDY Sleep Disturbance Ancillary Sub-Study - Patients undergoing surgery for valvular heart disease (VHD) are at high risk for adverse events, including high rates of post-operative delirium (POD). Should circadian disruption be found to be an important predictor in this high-risk population, safe, low cost, and easy to administer therapies to regulate circadian rhythm such as light therapy could be evaluated in future studies

The aims of this ancillary sub-study include:

1. To investigate the association between short sleep duration, less sleep regularity, and greater circadian rhythm disruption prior to surgery and POD within 7 days of VHD surgery.
2. To investigate the association between short sleep duration, less sleep regularity and greater circadian rhythm disruption (reduced melatonin and cortisol amplitudes) after surgery and POD within 7 days of VHD surgery.

Approximately 300 EMPRO trial participants will be enrolled into the ancillary study. The study is being conducted in highly experienced clinical centers in the U.S. and Canada. The estimated enrollment period is 12-15 months.

All eligible and consented patients in the parent EMPRO trial will be offered enrollment in this ancillary study through the parent trial consent process.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Planned de novo or redo:

  * Surgical aortic valve replacement SAVR ± ascending aortic repair (if circulatory arrest is not required) ± CABG
  * Mitral valve replacement (MVR) ± CABG
  * Mitral Valve Repair + CABG,
  * Double/Triple valve surgery ± CABG; Ross procedure These procedures can be done via a full or minimal-access sternotomy (using central aortic perfusion cannulae) with legally marketed valve(s), and can be done in combination with an left atrial appendage (LAA) closure/excision or partial/complete Maze procedure.
  * Valve sparing aortic root replacement (David procedure)
  * Valve sparing aortic root replacement (David procedure)
* No evidence of neurological impairment as defined by a NIHSS ≤1 and modified Rankin scale (mRS) ≤2 within 30 days prior to randomization
* Ability to provide informed consent and comply with the protocol

Exclusion Criteria:

* History of clinical stroke within 3 months prior to randomization
* Cerebral and or aortic arch arteriography or interventions within 3 days of the planned procedure
* Coronary catheterization within 3 days of index procedure, and the required repeat NIHSS score post-catheterization is worse than the screening/baseline NIHSS score conducted prior to the catheterization
* Active endocarditis at time of randomization with vegetation criteria
* Clinical signs of cardiogenic shock or treatment with IV inotropic therapy prior to randomization
* Participation in an interventional (drug or device) trial
* Isolated mitral valve repair, isolated tricuspid valve repair or combined mitral valve repair and tricuspid valve repair
* Anticipated requirement for prolonged mechanical ventilation greater than 48 hours after surgery in the opinion of the investigator
* Planned concomitant carotid endarterectomy during index surgical procedure

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 842 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who experience ischemic stroke and Acute Kidney Injury (AKI) | within 3 days post-randomization
  The combined number of patients who experience clinical ischemic strokes and acute kidney injuries that have occurred within 3 days post-randomization.
Number of patients who experience of death and delirium | by 7 days post-randomization
  The combined number of patients who experience death and delirium by 7 days post-randomization (with a blanking period for delirium of days 1 and 2 post-operatively).

SECONDARY OUTCOMES:
Proportion of patients who experience a clinical ischemic stroke | within 3 days post-randomization
  The proportion of patients who experience a clinical ischemic stroke within 3 days will be compared between the two groups (i.e., standard cannula versus the CardioGard device).
Proportion of patients who experience a clinical ischemic stroke | within 7 days post-randomization
  The proportion of patients who experience a clinical ischemic stroke within 7 days will be compared between the two groups (i.e., standard cannula versus the CardioGard device).
Number of patients with disabling clinical stroke | within 3 days post-randomization
  Number of patients with disabling clinical stroke within 3 days post-randomization
Number of patients with disabling clinical stroke | within 7 days post-randomization
  Number of patients with disabling clinical stroke within 7 days post-randomization
Neurological outcomes assessed by National Institutes of Health Stroke Scale (NIHSS) | within 3 days post-randomization
  Neurological outcomes are assessed by National Institutes of Health stroke Scale (NIHSS) to compare the treatment outcomes of three types of service delivery models. The NIHSS is an 11-item impairment scale to evaluate neurologic outcome and degree of recovery.
  Each item is scored between 0 and up to 4, total score ranges 0 (normal function) and a maximum possible score 42, with higher score indicating higher level of impairment.
  These assessments will be administered by blinded neurology trainees or study coordinators who are certified to administer the assessments.
Neurological outcomes assessed by National Institutes of Health Stroke Scale (NIHSS) | within 7 days post-randomization
  Neurological outcomes are assessed by National Institutes of Health stroke Scale (NIHSS) to compare the treatment outcomes of three types of service delivery models. The NIHSS is an 11-item impairment scale to evaluate neurologic outcome and degree of recovery.
  Each item is scored between 0 and up to 4, total score ranges 0 (normal function) and a maximum possible score 42, with higher score indicating higher level of impairment.
  These assessments will be administered by blinded neurology trainees or study coordinators who are certified to administer the assessments.
Number of patients with disabling clinical stroke determined by modified Rankin Scale (mRS) score ≥2 | at baseline
  Number of patients with disabling clinical stroke as indicated by mRS score ≥2. mRS will be assessed at baseline days.
  The scale runs from 0-6, running from perfect health without symptoms to death. A higher score indicates greater impairment.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to walk and attend own bodily needs without assistance.
  5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6 - Dead.
Number of patients with disabling clinical stroke determined by modified Rankin Scale (mRS) score ≥2 | at 30 days
  Number of patients with disabling clinical stroke as indicated by mRS score ≥2. mRS will be assessed at 30 days.
  The scale runs from 0-6, running from perfect health without symptoms to death. A higher score indicates greater impairment.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to walk and attend own bodily needs without assistance.
  5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6 - Dead.
Number of patients with disabling clinical stroke determined by modified Rankin Scale (mRS) score ≥2 | at 90 days
  Number of patients with disabling clinical stroke as indicated by mRS score ≥2. mRS will be assessed at 90 days.
  The scale runs from 0-6, running from perfect health without symptoms to death. A higher score indicates greater impairment.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to walk and attend own bodily needs without assistance.
  5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6 - Dead.
Montreal Cognitive Assessment (MoCA) Score | at baseline
  Global cognitive screening performance will be compared between groups and collected via the Montreal Cognitive Assessment (MoCA) - blind version at presurgical baseline.
  The MoCA scale is used for detecting cognitive impairment. The scores range between 0 to 30 points; a score of 26 or above was considered normal. Higher values represent a better outcome.
Montreal Cognitive Assessment (MoCA) Score | at 90 days
  Global cognitive screening performance will be compared between groups and collected via the Montreal Cognitive Assessment (MoCA) - blind version at 90 days.
  The MoCA scale is used for detecting cognitive impairment. The scores range between 0 to 30 points; a score of 26 or above is considered normal. Higher values represent a better outcome.
Montreal Cognitive Assessment (MoCA) Score | at 12 months
  Global cognitive screening performance will be compared between groups and collected via the Montreal Cognitive Assessment (MoCA) - blind version at 12 months.
  The MoCA scale is used for detecting cognitive impairment. The scores range between 0 to 30 points; a score of 26 or above is considered normal. Higher values represent a better outcome.
Oral Trail Making Test - Parts A and B (executive function) | at baseline
  The Trail Making Test consists of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). The patient should be instructed to connect the circles as quickly as possible, without lifting the pen or pencil from the paper. Time the patient connects the "trail." If the patient makes an error, point it out immediately and allow the patient to correct it. Results for part B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
Oral Trail Making Test - Parts A and B (executive function) | at 90 days post-randomization
  The Trail Making Test consists of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). The patient should be instructed to connect the circles as quickly as possible, without lifting the pen or pencil from the paper. Time the patient connects the "trail." If the patient makes an error, point it out immediately and allow the patient to correct it. Results for part B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
Oral Trail Making Test - Parts A and B (executive function) | at 12 months post-randomization
  The trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). The patient should be instructed to connect the circles as quickly as possible, without lifting the pen or pencil from the paper. Time the patient connects the "trail." If the patient makes an error, point it out immediately and allow the patient to correct it. Results for part B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
Wechsler Adult Intelligence Scale-Revised (WAIS-R) Digit Span (auditory-verbal attention) | baseline
  The WAIS-R Digit Span test assesses short term or working memory. The examinee listens to sequences of numbers orally and then repeats them as heard, in increasing order, and in reverse order. The raw scores for "digit span" range from a minimum of 2 to a maximum of 8. For this test, the longer the span the better the cognition; therefore, the higher score is the better outcome.
Wechsler Adult Intelligence Scale-Revised (WAIS-R) Digit Span (auditory-verbal attention) | at 90 days post-randomization
  The WAIS-R Digit Span test assesses short term or working memory. The examinee listens to sequences of numbers orally and then repeats them as heard, in increasing order, and in reverse order. The raw scores for "digit span" range from a minimum of 2 to a maximum of 8. For this test, the longer the span the better the cognition; therefore, the higher score is the better outcome.
Wechsler Adult Intelligence Scale-Revised (WAIS-R) Digit Span (auditory-verbal attention) | at 12 months post-randomization
  The WAIS-R Digit Span test assesses short term or working memory. The examinee listens to sequences of numbers orally and then repeats them as heard, in increasing order, and in reverse order. The raw scores for "digit span" range from a minimum of 2 to a maximum of 8. For this test, the longer the span the better the cognition; therefore, the higher score is the better outcome.
Wechsler Adult Intelligence Scale-Revised (WAIS-R) Digit Symbol Substitution Test (processing speed) | at baseline
  The WAIS-R Digit Symbol Substitution Test (DSST) is a paper-and-pencil cognitive test that consist of number-symbol pairs. It requires the examinee to copy, into spaces below rows of numbers, the symbols that are paired to each number. The DSST score is the number of digits coded correctly in a 90-second test period
Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test (verbal fluency/executive function) | at baseline
  The D-KEFS Verbal Fluency Test is comprised of three testing conditions: Letter Fluency, Category Fluency, and Category Switching. This test measures multiple aspects of verbal productivity and cognitive flexibility. It evaluates effectiveness of novel and semantic search strategies, and assesses flexibility in the implementation of word search strategies. There are three conditions in the test in which the examinee must say as many words as they can by letter, category, and category switching prompts.
Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test (verbal fluency/executive function) | at 90 days post-randomization
  The D-KEFS Verbal Fluency Test is comprised of three testing conditions: Letter Fluency, Category Fluency, and Category Switching. This test measures multiple aspects of verbal productivity and cognitive flexibility. It evaluates effectiveness of novel and semantic search strategies, and assesses flexibility in the implementation of word search strategies. There are three conditions in the test in which the examinee must say as many words as they can by letter, category, and category switching prompts.
Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test (verbal fluency/executive function) | at 12 months post-randomization
  The D-KEFS Verbal Fluency Test is comprised of three testing conditions: Letter Fluency, Category Fluency, and Category Switching. This test measures multiple aspects of verbal productivity and cognitive flexibility. It evaluates effectiveness of novel and semantic search strategies, and assesses flexibility in the implementation of word search strategies. There are three conditions in the test in which the examinee must say as many words as they can by letter, category, and category switching prompts.
Incidence of Delirium | first 7 days post-randomization
  The incidence of delirium will be assessed daily by the Confusion Assessment Method (3D-CAM or CAM-ICU) scale, or by the presence of a delirium adverse event, during the first 7 days post-randomization.
  The CAM consists of 4 features: 1-Onset, 2-Inattention, 3-Disorganized thinking, and 4-altered level of consciousness. The diagnosis of delirium by CAM is based on the presence of features 1 and 2, and either 3 or 4 and involves the presence/absence of delirium, but not its severity. Any error or behavioral observation consistent with a delirium feature means that feature is present.
Duration of Delirium | first 7 days post-randomization
  The duration of delirium will be measured as the number of days with positive CAM assessments or delirium adverse events by 7 days post-randomization.
  The CAM consists of 4 features: 1-Onset, 2-Inattention, 3-Disorganized thinking, and 4-altered level of consciousness. The diagnosis of delirium by CAM is based on the presence of features 1 and 2, and either 3 or 4.
Severity of Delirium | first 7 days post-randomization
  The severity of delirium will be measured during daily screening using standardized algorithms for extracting symptom severity from the 3D-CAM and CAM-ICU.
Number of Patients who experience Acute kidney injury (AKI) | within -7 days post-randomization
  Number of Patients who experience Acute kidney injury will be assessed within 7 days post-randomization.
All-cause mortality | within 90 days post-randomization
  All-cause mortality within 90 days post-randomization will be assessed.
All-cause mortality | within 12 months post-randomization
  All-cause mortality within 12-months post-randomization will be assessed.
Length of Index Hospitalization | at hospital discharge, up to 30 days
  Overall length of stay for the index hospitalization post-randomization will be measured and broken down by days spent in the ICU versus days not in the ICU.
Discharge disposition | at hospital discharge, up to 30 days
  Discharge disposition
Readmissions rates | first 90 days
  Readmission rates will be calculated for the first 90 days following randomization. Hospitalizations will be classified for all causes including for cardiovascular readmissions.
Readmissions rates | up to 1 year post-randomization
  Readmission rates will be calculated for the duration of follow-up, out to 1 year. Hospitalizations will be classified for all causes including for cardiovascular readmissions.
Days Alive out of Hospital | within 90 days post-randomization
  Days alive out of hospital and nursing/rehab facilities within 90 days after randomization
Actigraphy | 7-day period prior to index surgical procedure and Day 1 post index surgical procedure through hospital discharge
  Actigraphy data will be collected for a period of 7 days prior to the index surgical procedure. Actigraphic monitoring employs an accelerometer the size of a watch, which each study patient will wear on the wrist.
  Collected for participants in substudy.
Amount of Circadian Light | 7-day period prior to index surgical procedure
  A Speck light meter will be worn as a pendant while awake for a period of 7 days prior to surgery. Light measurements from light meters used as pendants are the closest to light measurements at eye level. The light meter will also be used to monitor the total amount of circadian light received by the patient.
  Collected for participants in substudy.
Photopic Light Levels | 7-day period prior to index surgical procedure
  A Speck light meter will be worn as a pendant while awake for a period of 7 days prior to surgery. Light measurements from light meters used as pendants are the closest to light measurements at eye level. The light meter will also be used to calculate photopic light levels
  Collected for participants in substudy.
Circadian Stimulus Values | 7-day period prior to index surgical procedure
  A Speck light meter will be worn as a pendant while awake for a period of 7 days prior to surgery. Light measurements from light meters used as pendants are the closest to light measurements at eye level. The light meter will also be used to calculate circadian stimulus values,
  Collected for participants in substudy.
Richards-Campbell Sleep Questionnaire | Day 1 post index surgical procedure through patient discharge from the ICU (average ICU stay is 3 days)
  Patients who are able to do so will be asked to fill out the Richards-Campbell Sleep Questionnaire (RCSQ), which is a brief 2-minute questionnaire designed for patient use in the ICU. Full score range from 0-100, with higher score indicating better sleep.
  Collected for participants in substudy.

CONTACTS AND LOCATIONS:
Overall Officials: Annetine C. Gelijns, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Steve Messe, MD, Principal Investigator — University of Pennsylvania; Alexander Iribarne, MD, Principal Investigator — Northwell Health
Locations (28):
- United States (24):
  - CHI St. Vincent Heart Institute, North Little Rock, Arkansas
  - Keck Hospital of the University of Southern California, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Bloomington, Indiana
  - Indiana Ohio Heart, Fort Wayne, Indiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins Medicine, Baltimore, Maryland
  - University of Maryland, College Park, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Columbia University Medical Center, New York, New York
  - New York Presbyterian-Cornell Medical Center, New York, New York
  - NYU Langone Hospital Brooklyn, New York, New York
  - Northwell Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - University Hospitals, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia
- Canada (4):
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hôpital Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified study data sets must be submitted to the designated NHLBI Program Official no later than 3 years after the end of the clinical activity (final patient follow-up, etc.) or 2 years after the main paper of the trial has been published, whichever comes first. Data are prepared by the study coordinating center and sent to the designated PO for review prior to release.
Access Criteria: Anyone who wishes to access the data. Any purpose. Data are available indefinitely at (Link to be included in the URL field below).
URL: https://biolincc.nhlbi.nih.gov/studies/